CLINICAL TRIAL: NCT03364829
Title: Utilizing Wearable Device to Observe the Clinical Response of COPD Patients Treated With Combined Bronchodilator and Home-based Pulmonary Rehabilitation Program
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Kuan Yuan Chen, Attending Physician of pulmonary medicine, Taipei Medical University Shuang Ho Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-JIRB Form057/20140202
Record Dates: First submitted 2017-11-11; First posted 2017-12-07 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: single group with comparisom before and after intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COPD on Indacaterol/Glycopyrronium (Experimental): COPD on indacaterol/glycopyrronium for 1 month
  Interventions: Drug: Indacaterol/Glycopyrronium

INTERVENTIONS:
Drug: Indacaterol/Glycopyrronium

SUMMARY:
The effectiveness of combined bronchodilator and exercise training on improving exercise capacity has been reported in COPD. However, little is known about effect of respective treatment in a real-time monitoring. Investigators applied wearable devices in monitoring continuously in COPD patients under treatment of combined dual bronchodilator and exercise training and research on associated inflammatory biomarkers profiles change

DETAILED DESCRIPTION:
The prevalence of chronic obstructive pulmonary disease (COPD) has increased year by year and the estimated mortality rate by 2030 will be in the fourth place. Estimated global prevalence of COPD in the population over age 40 is about 9-10% of the population. In Taiwan, the prevalence is about 16%. COPD is characteristic of irreversible airflow obstruction due to the pathological changes in the small airways, lung parenchyma and pulmonary vessels with chronic inflammation of the specific immune cells, as well as structural changes.

Although studies have suggested that exercise training in patients with COPD benefit the physical activity, but the anti-inflammatory benefits is unknown.Consider individual needs, this study will use the home mobile coach from Dr. Liu domestic development program to further investigate chronic obstructive pulmonary disease patients after receiving this training program,performance and analysis in the clinical laboratory to explore anti-inflammatory and pro-inflammatory between relevance and mechanisms in patients with COPD under real-time wearable devices monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Global Initiative for Chronic Obstructive Lung Disease (GOLD) according to diagnostic criteria of chronic obstructive pulmonary disease (age ≧ 40 years old and ≦ 85 years old), that the use of post-bronchodilator inhalation, pulmonary function test results of the forced expiratory volume first second (FEV1.0) / forced vital capacity (FVC) <70% 2. COPD patients is not currently accepting any pulmonary rehabilitation program 3. Currently in a stable condition, after researchers explained the purpose of this study, the researchers agreed to participate.

Exclusion Criteria:

1. Asthma, bronchiectasis, tuberculosis, pneumoconiosis, or other pulmonary diseases
2. Associated with neuromuscular function disorders such as hemiplegia or no independent walking function;
3. Severe heart disease, such as acute myocardial infarction, serious or heart failure, etc.
4. Diagnosed with severe mental disorders such as dementia or poor compliance
5. Acute exacerbation or infection in 3 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Combined dual bronchodilator and protocolized pulmonary rehabilitation effect on daily activity in step counts per 24 hours | Investigators would measured daily step counts for each patients at baseline, 1 month and 4th month after intervention
  Change from baseline daily activity in step counts per 24 hours at 1 month after dual bronchodilator therapy and at 4th month after further combined dual bronchodilator with protocolized pulmonary rehabilitation therapy for 3 months. Daily step counts measured by wearable devices was represented for daily activity
Combined dual bronchodilator and protocolized pulmonary rehabilitation effect on 6 minutes walking distance in meters | Investigators would measured daily steps for each patients at baseline, 1 month and 4th month after intervention
  Change from baseline 6 minutes walking distance in meters at 1 month after dual bronchodilator therapy and at 4th month after further combined dual bronchodilator with protocolized pulmonary rehabilitation therapy for 3 months.
Combined dual bronchodilator and protocolized pulmonary rehabilitation effect on heart rate variability | Investigators would measured heart rate variability in ratio of low frequency and high frequency for each patients at baseline, 1 month and 4th month after intervention
  Change from baseline heart rate variability in ratio of low frequency and high frequency at 1 month after dual bronchodilator therapy and at 4th month after further combined dual bronchodilator with protocolized pulmonary rehabilitation therapy for 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kang-Yuan Lee, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No